CLINICAL TRIAL: NCT04663724
Title: Computer-Based Treatment for Social Anxiety Disorder, A Randomized Controlled Trial
Brief Title: Computer - Based Treatment for Social Anxiety Disorder
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: In June 2023 NYSPI undertook an Institute-wide safety review of research protocols that involve human subjects. To support the safety review, NYSPI, paused all ongoing human subjects research studies as of June 12, 2023
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); Mclean Hospital (Other); Tel Aviv University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Franklin Schneier, Director, Anxiety Disorders Clinic, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8072; 5R33MH116089-04 (NIH)
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Social Anxiety Disorder
Keywords: Attention
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Computer-Based Treatment (Experimental): A 4-week (8-sessions) course of computer-based treatment. Participants will receive treatment twice a week for four weeks.
  Interventions: Behavioral: Computer-Based Treatment
- Comparator Computer-Based Treatment (Active Comparator): A 4-week (8-sessions) course of computer-based treatment. Participants will receive treatment twice a week for four weeks.
  Interventions: Behavioral: Computer-Based Treatment

INTERVENTIONS:
Behavioral: Computer-Based Treatment — A 4-week (8 30-minute sessions) course of computer-based treatment involving viewing pictures of faces while music may play. Participants will receive research treatment twice a week.

SUMMARY:
The present study is a controlled trial that seeks to examine the feasibility, acceptability, mechanism, and efficacy of a recently developed computer-based therapy in individuals with social anxiety disorder (SAD)

DETAILED DESCRIPTION:
This randomized clinical trial examines the feasibility, acceptability, mechanism, and relative efficacy of two forms of a recently developed 4-week/8-session computer-based therapy in individuals with social anxiety disorder (SAD). The purpose of this study is to assess whether a brief computer-based research treatment, provided in 30 minutes sessions, helps improve social anxiety symptoms, and by what mechanism. The study will also assess the effect of research treatments on brain activity using magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 to 60
* Current primary diagnosis of SAD
* Score of at least 50 on the Liebowitz Social Anxiety Scale (self-rated version)
* Fluent in English
* Willing and able to give informed written consent
* Ability to participate responsibly in the protocol
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Present or past psychotic episode, psychotic disorder, schizophrenia, schizoaffective disorder, or bipolar disorder
* Current severe depression
* Suicidal ideation or behavior
* Current diagnosis of post-traumatic stress disorder, obsessive-compulsive disorder, bipolar disorder, manic episode or tic disorder
* Current or past organic mental disorder, seizure disorder, epilepsy or brain injury
* Current unstable or untreated medical illness
* Severe alcohol use disorder, severe cannabis use disorder, and any severity of other substance use disorder (except nicotine use disorders)
* Use of psychiatric medication in the past month other than a stable dose of selective serotonin reuptake inhibitors (SSRIs) for at least 3 months
* Any concurrent cognitive behavioral therapy or other psychotherapy that was initiated in the past 3 months
* Pregnancy, or plans to become pregnant during the period of the study (will be assessed by urine)
* Contraindication to MRI scanning (Paramagnetic metallic implants or devices contraindicating magnetic resonance imaging or any other non-removable paramagnetic metal in the body)

  1. pacemaker
  2. paramagnetic metallic prosthesis
  3. surgical clips
  4. shrapnel
  5. necessity for constant medicinal patch
  6. some tattoos
* Inability to tolerate MRI scanning procedures (i.e., severe obesity, claustrophobia)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Total Score of Liebowitz Social Anxiety Scale (LSAS) | From baseline up to Month 4
  Clinician-rated scale scoring anxiety (0, none to 3, severe) and avoidance (0,none to 3, severe) in 24 social situations for a total score of 0 to 144. Higher scores indicate greater social anxiety.
Change in Total Score of Quality of Life Enjoyment & Satisfaction Questionnaire | From baseline up to Month 4
  Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q): self-rated assessment of quality of life. 16 items related to life quality, each rated on a score of 1 (very poor) to 5 (very good), with a minimum total score of 16, and a maximum total score of 80.

SECONDARY OUTCOMES:
Change in Total Score of Social Phobia Inventory (SPIN) | Baseline to Month 4
  The Social Phobia Inventory (SPIN) is a self-rated questionnaire used to assess severity of social anxiety disorder. 17 items related to social anxiety each rated on a score of 0 to 4, with a minimum total score of 0 (least social anxiety), and a maximum total score of 68 (most social anxiety).
Clinical Global Impression-Change Scale | Baseline to Month 4
  Clinical Global Impression-Change Scale: An observer rating of overall clinical change, with rating from 1 (very much improved) to 7 (very much worse). Responder category is defined by a score of 1 or 2.

CONTACTS AND LOCATIONS:
Overall Officials: FRANKLIN SCHNEIER, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the National Database for Clinical Trials related to Mental Illness (NDCT). We will obtain information needed to generate a Global Unique Identifier (GUID) for each participant (sex, first name, last name, middle name, date of birth, and city/municipality of birth). Raw data will be submitted semi-annually every January 15 and July 15, and prior to the end of each grant.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 12 months after completion of study assessments